CLINICAL TRIAL: NCT03614819
Title: Laser Used in the Treatment of Hypomineralized Occlusal Lesions in Teeth Enamel Affected by MIH: a Randomized Controlled Clinical Study
Brief Title: Laser Used in the Treatment of Hypomineralized Occlusal Lesions in Teeth Enamel Affected by MIH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Luciana Pion Antonio, Principal investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MIHForp
Record Dates: First submitted 2018-06-14; First posted 2018-08-03 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Dental Enamel Hypoplasia
Keywords: Lasers; Dental enamel hypoplasia; Preventive dentistry; Dental caries
MeSH Terms: conditions — Dental Enamel Hypoplasia; Dental Caries

STUDY DESIGN:
Intervention Model Description: Diode laser group Prophylaxis of the selected region for the study and application of diode laser (Sirolaser, Sirona Dental Systems GmbH, Bensheim, Germany) with wavelength of 970 nm +/- 10 nm, maximum power of 7 W CW, 1mW guide beam and 320μm optical fiber. Irradiation will be performed on the entire occlusal surface in contact mode, with power of 0.7 W and frequency of 10 Hz for 30 seconds, having an energy density of 222.82 J / cm2.
  Glass Ionomer Sealing Group Prophylaxis of the selected region for the study, followed by relative insulation with cotton rollers of the tooth in question, application of acid polyacrylic for 15 seconds throughout the surface, light drying with cotton ball, insertion of the high viscosity glass ionomer (Equia Forte in capsule - GC) through a specific applicator, after loss of the gloss of the digital pressure material with Vaseline for due drainage and surface protection of the material.
Masking Description: No masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Diode laser group (Experimental): Prophylaxis of the selected region for the study with Robson brush and prophylactic paste, washing and drying, followed by application of diode laser (Sirolaser, Sirona Dental Systems GmbH, Bensheim, Germany) with wavelength of 970 nm +/- 10 nm, maximum power of 7 W CW, 1mW guide beam and 320μm optical fiber. Irradiation will be performed on the entire occlusal surface in contact mode, with power of 0.7 W (energy of 70 mJ) and frequency of 10 Hz for 30 seconds, having an energy density of 222.82 J / cm2. The FieldMaxII-TOP power meter (Coherent, Inc, USA) will be used prior to and after the applications. The laser will be applied in a sweeping motion throughout the affected surface, the fiber being maintained positioned perpendicular to the occlusal surface throughout the movement. The irradiation time will be standardized in 30 seconds.
  Interventions: Procedure: Diode laser group
- Glass Ionomer Sealing Group (Active Comparator): Prophylaxis of the selected region for the study with Robson brush and prophylactic paste, washing and drying with cotton balls, followed by relative insulation with cotton rollers of the tooth in question, application of acid polyacrylic for 15 seconds throughout the surface, light drying with cotton ball, insertion of the high viscosity glass ionomer (Equia Forte in capsule - GC) through a specific applicator, after loss of the gloss of the digital pressure material with Vaseline for due drainage and surface protection of the material, removal of the excess, checking the occlusion with carbon paper, occlusal adjustments if necessary, superficial protection with petroleum jelly.
  Interventions: Procedure: Glass Ionomer Sealing Group

INTERVENTIONS:
Procedure: Diode laser group — Prophylaxis of the selected region for the study with Robson brush and prophylactic paste, washing and drying, followed by application of diode laser (Sirolaser, Sirona Dental Systems GmbH, Bensheim, Germany) with wavelength of 970 nm +/- 10 nm, maximum power of 7 W CW, 1mW guide beam and 320μm optical fiber. Irradiation will be performed on the entire occlusal surface in contact mode, with power of 0.7 W (energy of 70 mJ) and frequency of 10 Hz for 30 seconds, having an energy density of 222.82 J / cm2. The FieldMaxII-TOP power meter (Coherent, Inc, USA) will be used prior to and after the applications. The laser will be applied in a sweeping motion throughout the affected surface, the fiber being maintained positioned perpendicular to the occlusal surface throughout the movement. The irradiation time will be standardized in 30 seconds.
  Arms: Diode laser group
Procedure: Glass Ionomer Sealing Group — Prophylaxis of the selected region for the study with Robson brush and prophylactic paste, washing and drying with cotton balls, followed by relative insulation with cotton rollers of the tooth in question, application of acid polyacrylic for 15 seconds throughout the surface, light drying with cotton ball, insertion of the high viscosity glass ionomer (Equia Forte in capsule - GC) through a specific applicator, after loss of the gloss of the digital pressure material with Vaseline for due drainage and surface protection of the material, removal of the excess, checking the occlusion with carbon paper, occlusal adjustments if necessary, superficial protection with petroleum jelly.
  Arms: Glass Ionomer Sealing Group

SUMMARY:
Background: Nowadays an increase in the incidence of teeth affected by molar incisor hypomineralisation (MIH) has been observed. There are several treatment modalities that depend on the degree of severity of the defect, such as preventive procedures, restorative and even dental extractions. However, these changes may affect the retention and longevity of restorative materials. Therefore, the aim of this study is to evaluate the use of diode laser irradiation for the treatment of occlusal surfaces of moderate lesions in permanent first molars affected with MIH as a preventive method for dental caries and occlusal wear, besides verifying the discomfort of the treatment by patients. Methods: For this, a controlled and randomized study, with parallel groups, will be conducted comparing the treatment with diode laser and sealing with high viscosity glass ionomer cement in the teeth affected by the MIH. Participants will be assessed at baseline and after 1 week, 1, 6, 12, 18 and 24 months. As the main outcome, the presence of dentin caries lesion and /or occlusal surface wear included in the study with dentin involvement will be evaluated. A visual examination for caries detection will be done using the ICDAS, using the index based on classification in the United States Public Health Service - Modified (USPH) for evaluation of sealed teeth and impression of impacted teeth for quantitative analysis of the lesions. Other outcomes such as patient satisfaction with treatment, patient discomfort, impact on quality of life and participant perception, as well as the duration and cost of treatment, as well as their cost-efficacy, will also be evaluated. Multilevel statistical analyzes will be performed to verify the efficacy of Diode laser treatment compared to sealing, in addition to possible factors associated with this efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Children who present at the first permanent molar with occlusal surface affected with light or moderate severity of MIH
* Children between 6 and 10 years old

Exclusion Criteria:

* Teeth that present restorations
* Teeth that presente sealants
* Enamel malformations that are specific to some syndromes
* Hypomineralized enamel affected by the ingestion of fluoride during enamel development

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 122 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of clinical signs change in the progression of caries lesion and / or occlusal surface wear during the follow-up | All surfaces will be examined after previous cleaning with prophylactic paste and water and a Robson brush, with lighting and after air drying and 1, 6, 12, 18 and 24 months after
  The main outcome will be the presence of changes in clinical signs in relation to the progression of carious lesions and / or occlusal surface wear included in the study with dentin involvement through ICDAS, photographs, radiographic examination and the index based on the classification in the United States Public Health Service - Modified (USPH).

SECONDARY OUTCOMES:
Satisfaction in relation the treatment using VAS scale | This evaluation will be applied after 1 week of treatment, 1, 12 and 24 months and will not be identified by name and will be done in the absence of the operators so as not to restrain the subject from expressing their actual opinion.
  The responsibles will be asked to respond about the satisfaction regarding the care (treatment and follow-up) received by their children. He should classify his satisfaction using the VAS scale with indexes from 0 to 10, with 0 being the worst evaluation of treatment and 10 being the best.
Self-reported discomfort using Wong Backer face scale after the treatment | This evaluation will be performed before starting the treatment with laser or with high viscosity glass ionomer and 2 minutes after the treatment is performed]
  In order to assess the discomfort reported by the children in relation to the type of treatment received, the same timekeeping operator will apply the Wong-Baker Facial Scale to the patient, which is composed of six figures with equidistant faces that the first one is very smiling and the expressions are changing, until the last one is very sad. The face 1 mean "no hurts", face 2 "hurts little bit", face 3 "hurts little more", face 4 "hurts even more", face 5 "hurts whole lot", face 6 "hurts worst". The child chooses the face that judges more similar to his own after the treatment.
Hypersensitivity to dentin | This evaluation will be performed before treatment, 1 week, 1, 6, 12, 18 and 24 months after inclusion
  The patients will answer to a VAS scale with indexes from 0 to 10 (no pain - 0 and worst pain - 10) for each teeth.
Evaluation of patient's perception of satisfaction regarding their oral health | For this, an external examiner will apply the questionnaire prior to randomization and on 1, 12 and 24 month return visits.
  The evaluation of the patient's perception of satisfaction regarding his / her oral health will be performed through the questionnaire of quality of life, Child Perceptions Questionnaire 8-10 (CPQ8-10), specially developed for children aged 8-10 years old.
  The questionnaire consists of 10 questions. Each question is composed of 5 answers: a) Never, b) Once or twice, c) Sometimes, d) Often, e) Every day or almost every day. These issues include generic and specific aspects of oral diseases. For example: "In the last month, how many times have you had toothache or mouth pain?" or "In the last month, how many times have you felt sad because of your teeth or your mouth?"
Costs of each consultation performed through study completion | The time spent in each of the sessions will be timed by an external examiner not participating in the exams, who will also note the number of visits of each participant. The data will be collected at all return visits (1 week, 1, 6, 12, 18 and 24 months)
  To calculate the direct costs of the procedures, the time spent in each consultation (initials and reevaluations) will be taken into account. For the calculation of direct costs, the prices of consumer and permanent materials (specifications and quantity) used in each procedure, electricity and the professional fee will be considered.

CONTACTS AND LOCATIONS:
Locations (1):
- Luciana Pion Antonio, Ribeirão Preto, São Paulo, Brazil